CLINICAL TRIAL: NCT03187535
Title: The Effect of Transcutaneous Electric Acupoint Stimulation on Post-operative Nausea and Vomiting After Spinal Surgery
Brief Title: Effect of TEAS on PONV After Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jyoti Pandya (Other)
Responsible Party: Sponsor-Investigator, Jyoti Pandya, M.D., Principal Investigatgor, Associate Attending, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017H0101
Record Dates: First submitted 2017-05-15; First posted 2017-06-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: PONV
Keywords: Transcutaneous Electrical Acupoint Stimulation
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant will be blinded to the treatment arm; all investigators and care providers will be blinded to the treatment arm. Only the anesthesiologist trained in acupuncture and administering the treatment will know the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcutaneous Electrical Acupoint Stimulation (Experimental): Subjects in the "Transcutaneous Electrical Acupoint Stimulation" (TEAS) group will receive 20 minutes of TEAS via ES-130 beginning at the time ondansetron is administered (usually given 30 minutes before the end of surgery), for prevention of PONV.
  Interventions: Device: TEAS via ES-130
- No Transcutaneous Electrical Acupoint Stimulation (Sham Comparator): Subjects in the "No Transcutaneous Electrical Acupoint Stimulation" group will not receive any TEAS, although they will have the acupoints identified and ECG patches placed. The device will not be connected to the electrodes of the ES-130 device at the end of surgery, and no TEAS will be delivered.
  Interventions: Other: No TEAS

INTERVENTIONS:
Device: TEAS via ES-130 — Transcutaneous Electrical Acupoint Stimulation will be administered delivered by the ES-130 device for 20 minutes at the time ondansetron is given (typically 30 minutes before the end of surgery). Subjects randomized to this intervention will have the TEAS device connected to the previously placed ECG patches to deliver the stimulus.
  Arms: Transcutaneous Electrical Acupoint Stimulation
Other: No TEAS — No Transcutaneous Electrical Acupoint Stimulation will be delivered to the subjects randomized to this group; ECG patches will be placed at the identified acupoints, however, no electrical stimulus will be delivered.
  Arms: No Transcutaneous Electrical Acupoint Stimulation

SUMMARY:
The proposed research will utilize electroacupuncture, a type of needleless acupuncture that uses electrostimulation, in a randomized, double blind study, to evaluate the incidence of post-operative nausea and vomiting (PONV) in patients undergoing spinal surgeries with the transcutaneous electrical acupoint stimulation (TEAS) compared to patients without TEAS.

DETAILED DESCRIPTION:
The rates of PONV will be evaluated over the first 24 hours after surgery, opioid consumption in units of morphine equivalence, and any adverse side effects will be recorded. Subjects who are included in the research will be randomly assigned to one of two groups - one group is the control group, receiving no TEAS, and the other group receiving TEAS. An anesthesiologist trained in acupuncture will utilize the Excel Pointer to locate the specific acupoints previously identified as associated with prevention PONV. Anesthesiologist will place electrocardiogram (ECG) pads at the identified acupoints prior to surgery. Subjects will be connected to the ES-130 (electro-therapy) device upon entering the operating room. Prior to the surgical closure, the unblinded researcher will initiate delivery of TEAS, or not, according to study protocol based on the randomization group of the participant. The anesthesiologist will not know the group assignment. At the end of surgery, the subject will be disconnected from the ES-130 and the ECG pads will be carefully removed. Researchers will follow up with the subject in recovery regarding any occurrence and severity of PONV, adverse events, and verbal pain scores, until 24 hours after end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients , 18 or older
* American Society of Anesthesiologists (ASA) classification I or II or III
* Undergoing elective spinal surgery expected to last no more than four hours (from induction of anesthesia to extubation).
* Capable and willing to consent

Exclusion Criteria:

* Neuraxial (intrathecal or epidural) block
* Significant ongoing history of vestibular disease or dizziness
* Nausea or vomiting within 24 hours prior to surgery, use of antiemetic or emetogenic drugs within 3 days of surgery
* Documented alcohol or substance abuse within 3 months before the surgery
* Limb abnormalities such as burn and amputation.
* Poorly controlled diabetes mellitus (fasting plasma glucose >126 mg/dL or <70 mg/dL)
* Implantation of metal/electrical devices, such as nerve stimulator, cardiac pacemaker, cardioverter, defibrillator and internal hearing aids
* Rash, local infection, keloid, any dermatologic condition that could interfere with the acupoint stimulation area
* Documented alcohol or substance abuse within 3 months before surgery
* Presence of clinically diagnosed major psychiatric condition such as bipolar disorder, uncontrolled major depression, or schizophrenia
* Chemotherapy or radiation therapy within 7 days before surgery
* Investigational product use within 3 months prior surgery
* Any condition, which in the opinion of the investigator would make subject ineligible for participation in the study (history of unstable cardiovascular, pulmonary, renal, hepatic, seizures)
* Special population (prisoners, pregnant and lactating women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
incidence of PONV | up to 24 hours after surgery
  measure the incidence of PONV in spinal surgery
severity of PONV | up to 24 hours after surgery
  use Verbal Rating Scale (VRS) score (0-10) to rate nausea

SECONDARY OUTCOMES:
Time to first nausea/vomiting rescue medication | within 2 and 24 hours after surgery
  Time until subject requests rescue anti-emetic therapy
opioid consumption (units of morphine equivalence) | 2 and 24 hours after surgery
  compare the opioid consumption after surgery in units of morphine
incidence of adverse events | 24 hours after surgery
  compare incidence of adverse events between groups

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bergese, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No